CLINICAL TRIAL: NCT00483899
Title: Double-blind, Placebo-controlled, 3-way Crossover Study to Investigate the Effect of 7-days Repeat Once Daily Inhaled Doses of GW870086X Administered Via DISKHALER on Airway Responsiveness to AMP in Mild Steroid-naive Male Asthmatics
Brief Title: Examine the Effect of Repeat Inhaled Doses of GW870086X on Lung Function in Mild Asthmatic Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SIG102335
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: GW870086X Asthma Crossover repeat dose inhaled
MeSH Terms: conditions — Asthma | interventions — GW870086X

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: Part A (Experimental): Subjects in Cohort 1 will be randomized to receive 0.5, 2 and 6 mg GW870086X and placebo.
  Interventions: Drug: GW870086X; Drug: Placebo
- Cohort 2: Part A (Experimental): Subjects in Cohort 2 will be randomized to receive 3 mg GW870086X or placebo.
  Interventions: Drug: GW870086X; Drug: Placebo
- Part B (Experimental): Subjects will be randomized to receive 1 and 3 mg of GW870086X or placebo.
  Interventions: Drug: GW870086X; Drug: Placebo

INTERVENTIONS:
Drug: GW870086X — Subjects will inhale 0.25 or 1.5 mg/inhalation GW870086X for four times
Drug: Placebo — Placebo matching GW870086X will be administered by subjects

SUMMARY:
This study was designed to look at safety aspects and effects of repeat inhaled doses of GW870086X in mild asthmatics to develop this drug for its use in asthma and chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion criteria:

* Male subjects aged 18-55
* Documented history of bronchial asthma diagnosed at least 6 months ago.
* Only being treated with short-acting beta-2-agonist therapy e.g. Ventolin
* Documented sensitivity to adenosine mono phosphate (AMP) at screening visit
* Demonstrate repeatable and reproducable response to inhaled AMP at the run-in visit

Exclusion criteria:

* Any significant illness or disease
* History of life threatening asthma
* History of respiratory tract infection
* Subjects who take medication for their asthma, or other conditions, not compatible with this study.
* Smoker
* Subjects who are oversensitive to corticosteroids
* History of drug or alcohol abuse
* Donated blood within last 3 months
* Been involved in another clinical trial during the last 3 months
* Subjects who work night shifts
* Subjects who are undergoing de-sensitisation therapy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-10-07 (Actual); Primary Completion 2006-12-15 (Actual); Study Completion 2006-12-15 (Actual)

PRIMARY OUTCOMES:
Change in lung function 2 hours after treatment on day 7 | on day 7

SECONDARY OUTCOMES:
Change in lung function 14 and 26 hours after treatment on day 7; Change in lung function 2 hours after treatment on day 1; Effects on blood and urine tests; effects on the heart, pulse rate and blood pressure; effects on the lungs | 2 hours after treatment on day 1, 14 and 26 hours after treatment on day 7;

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, London

REFERENCES:
- See also: Results for study SIG102335 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/SIG102335?search=study&search_terms=SIG102335#rs